CLINICAL TRIAL: NCT05027581
Title: A Phase IIb Study to Evaluate the Efficacy and Safety of Chondrochymal® for Subjects With Knee Osteoarthritis (Knee OA)
Brief Title: Chondrochymal® for Subjects With Knee Osteoarthritis (Knee OA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiwan Bio Therapeutics Inc. (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chondrochymal-01
Record Dates: First submitted 2021-08-19; First posted 2021-08-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Knee
Keywords: knee osteoarthritis; BM-MSC
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chondrochymal® group (Experimental): Subjects will be IA injected at the target knee with 3 mL of Chondrochymal® containing 5.0 x 107 BM-MSCs in lactated Ringer's solution at Day 1.
  Interventions: Drug: Bone marrow mesenchymal stem cells
- Hya-Joint Plus Synovial Fluid Supplement (Active Comparator): Hya-Joint Plus Synovial Fluid Supplement containing 60 mg/3 mL of hyaluronic acid will be IA administrated into the subject's target knee at Day 1.
  Interventions: Drug: hyaluronic acid

INTERVENTIONS:
Drug: Bone marrow mesenchymal stem cells — The bone marrow mesenchymal stem cells (BM-MSCs) in Chondrochymal® for this study was obtained from the donor recruited in Taipei Veterans General Hospital, Taiwan. Donors aged 20 to 50 and tested negative to infection of human immunodeficiency virus type 1 and 2 (HIV-1/2), hepatitis B virus (HBV), hepatitis C virus (HCV), Cytomegalovirus (CMV), Treponema pallidum (syphilis), human T-lymphotropic virus types I and II (HTLV-I/II), and Tuberculosis (TB) were enrolled. The eligible donor's bone marrow was aspirated from the iliac crest or femur. The collected BM-MSCs were then cultured, expanded and cryopreserved in a Good Tissue Practice (GTP)-complied laboratory. The qualified cells in cryopreservation meeting the release criteria will be thawed, mixed with lactated Ringer's solution, and transferred into a sterile syringe as the final product.
  Other Names: Chondrochymal®
  Arms: Chondrochymal® group
Drug: hyaluronic acid — (60 mg/3 mL hyaluronic acid [HA])
  Other Names: Hya-Joint Plus Synovial Fluid Supplement
  Arms: Hya-Joint Plus Synovial Fluid Supplement

SUMMARY:
This is a randomized, single-blind, parallel, active-controlled study to evaluate the efficacy and safety of bone marrow mesenchymal stem cells (BM-MSCs), Chondrochymal®, in subjects aged 40 to 80 with knee OA.

DETAILED DESCRIPTION:
This phase IIb study is a prospective, single-blind, parallel, active-controlled study to evaluate the efficacy and safety of Chondrochymal® in subjects with knee OA. All the subjects will be enrolled in Taiwan. The target population is composed of subjects with unilateral or bilateral OA knee(s). For subjects with bilateral OA knees, only the knee with more severe symptoms will be selected as the target knee. If the severities of the OA symptoms are the same for both knees, the knee with more pain should be selected, where the WOMAC pain score will take the priority over the VAS index. Eligible subjects will be randomized into one of the study groups, Chondrochymal® Group or Control Group, in 1:1 ratio. To keep the blindness, the subject's eyesight will be masked by a curtain while receiving the IA injection.

ELIGIBILITY:
Inclusion Criteria:

1. All genders aged 40 to 80 (inclusive).
2. WOMAC pain score equals to or higher than 7 in the target knee.
3. Subject with unilateral/bilateral OA knee(s) of Kellgren-Lawrence grading II-IV, who is not suitable for or unwilling to undergo knee surgery (including total knee replacement).
4. Pain of the target knee as assessed by Visual Analogue Scale (VAS) equals to or higher than 4.
5. Body mass index (BMI) between 20 and 35 kg/m2.
6. Has received conventional therapies for knee OA (e.g., analgesic administration or physical therapy) for more than 3 months but the symptoms have not relieved.
7. With adequate hematological indices: - White blood cell (WBC) ≥ 3,000/mm3 - Platelet count ≥ 80,000/μL - Prothrombin time (PT), international normalized ratio (INR), and activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of the normal range (ULN)
8. With adequate liver function where serum total bilirubin ≤ 1.5 times ULN, aspartate aminotransferase (AST) ≤ 3 times ULN, and alanine aminotransferase (ALT) ≤ 3 times ULN.
9. Has an estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m2, calculated by the Modification of Diet in Renal Disease (MDRD) equation.
10. Understand and sign the informed consent form.

Exclusion Criteria:

1. With congenital or acquired bone hypoplasia (Varus more than 10° or Valgus more than 20°).
2. Had any intra-articular (IA) injection or surgery of the target knee within 3 months prior to screening, or had received any prior cell therapy on the target knee.
3. With severe knee osteoarthritis on the target knee who has decided to receive surgery (including total knee replacement) per surgeon's advice before screening.
4. With coagulation or hematological disorder not suitable for IA injection.
5. Administered or requiring systemic or topical on the target knee joint immunosuppressive agent, anti-inflammatory drug, steroid, analgesics, opioid, or duloxetine for knee OA, except for acetaminophen (oral daily dose ≤ 2000 mg or topical use at any dose level), Etoricoxib (oral daily dose ≤ 120 mg or topical use at any dose level), and Celebrex (oral daily dose ≤ 200 mg or topical use at any dose level), within 1 week prior to screening. For long-acting steroids (e.g., dexamethasone), a subject received systemic treatment within 2 weeks before screening will be excluded. A subject requiring routine use of low-dose Aspirin for preventing thrombosis (≤ 100 mg/day) will not be excluded from this study.
6. With spontaneous knee osteonecrosis on either knee.
7. With crippled lower limb(s) rated ACR functional class IV (Largely or Wholly Incapacitated) or cannot walk without one/two arm(s)-operated walking assisting device (defined by CNS15390).
8. With effusion, bleeding, ligament instability, arthrochalasis, muscular or neurological diseases causing deformity of the knee joint, or any joint diseases other than OA on the target knee.
9. Active systemic infection or acute infection around the target knee joint.
10. Any significant dermatological disease near the injection site that is not suitable for IA injection at the investigator's discretion.
11. Has claustrophobia and/or cannot take magnetic resonance imaging (MRI) test.
12. Any metal devices placed in the body such as pacemaker, artificial heart valve, or hemostatic clamps/clips for intracranial aneurysm posing risk under magnetic field (of MRI).
13. Previous surgery of the target knee that may cause metal imaging artifacts on imaging study.
14. Known or possible allergy to components of the study drugs or rescue medications.
15. Any form of primary immunodeficiency or autoimmune disease requiring systemic immunosuppressive therapy.
16. Subjects with malignant tumors or benign tumors that may interfere with the study treatment or subsequent evaluation.
17. Has serious medical conditions such as renal (estimated glomerular filtration rate < 30 mL/min/1.73m2), hepatic (e.g., Child-Pugh Class C), psychiatric condition (e.g., alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the subject.
18. Currently with confirmed or suspected active infection of HIV, HBV, or HCV at the investigator's discretion.
19. Has received cytotoxic agent, chemotherapy, or radiotherapy that could interfere with the efficacy of investigational product within 3 months of the screening visit.
20. Had prior investigational therapy (including cell therapy) within the past 3 months prior to subject's Screening Visit.
21. Female subject of childbearing potential who:

    * Is lactating; or
    * Has positive pregnancy test result at eligibility checking; or
    * Refuses to adopt at least one form of birth control from signing informed consent to the end of the study.
22. Male subject with female spouse/partner who is of childbearing potential refuses to adopt at least one form of birth control from signing informed consent to the end of the study. For exclusion criteria #21 and #22, acceptable forms of birth control include:

    * Established use of oral, injected or implanted hormonal methods of contraception.
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps).
23. Physiologically or psychologically inappropriate for participating in the study per investigator's judgment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Efficacy-Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) assessment | Week 24
  Change from baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score on the target knee at Week 24.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC LK 3.1) is applied extensively to patients with osteoarthritis of the hip or knee. It is a 24-item patient-reported questionnaire with a total score ranging from 0 to 96. The sub-scores range from 0 to 4 for each item with a higher score indicating a more severe OA symptom. The WOMAC includes 3 domains: (1) Pain: 5 items (score range: 0 to 20), (2) Stiffness: 2 items (score range: 0 to 8), and (3) Functional limitation: 17 items (score range: 0 to 68).
  For ease of interpretation, WOMAC scores (including total scores and sub-scores) will be linearly transformed to a 0 to 100 scale.

SECONDARY OUTCOMES:
Efficacy-Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) assessment | Week 4、Week 12、Week 24、Week 36、Week 52
  Change from baseline at each post-treatment visit during the Evaluation Period on the target knee in total scores and sub-scores of each section of WOMAC.
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC LK 3.1) is applied extensively to patients with osteoarthritis of the hip or knee. It is a 24-item patient-reported questionnaire with a total score ranging from 0 to 96. The sub-scores range from 0 to 4 for each item with a higher score indicating a more severe OA symptom. The WOMAC includes 3 domains: (1) Pain: 5 items (score range: 0 to 20), (2) Stiffness: 2 items (score range: 0 to 8), and (3) Functional limitation: 17 items (score range: 0 to 68).
  For ease of interpretation, WOMAC scores (including total scores and sub-scores) will be linearly transformed to a 0 to 100 scale.
Efficacy-Visual Analogue Scale (VAS) assessment | Week 4、Week 12、Week 24、Week 36、Week 52
  Change from baseline at each post-treatment visit during the Evaluation Period on the target knee in the Visual Analogue Scale (VAS) for pain.
  The Visual analog scale (VAS) pain assessment measures pain intensity. It is a scale of 10 cm in length, representing the subject's pain intensity with higher scores indicating more severe pain. VAS score ranges from 0 to 10 cm, and will be transformed to a "0 to 100" mm scale.
Efficacy-SF-36 Quality of Life (QoL) health survey questionnaire | Week 4、Week 12、Week 24、Week 36、Week 52
  Change from baseline at each post-treatment visit during the Evaluation Period in the domain scores and total score of SF-36 Quality of Life (QoL) health survey questionnaire.
  The SF-36 Quality of Life (QoL) health survey questionnaire (v2.0) is a standardized, self-evaluated measurement of health status. It has 36 questions to measure functional health and well-being from the patient's point of view. The SF-36 QoL questionnaire consists of 8 scaled scores in various health domains including 4 items in vitality, 10 items in physical functioning, 2 items in bodily pain, 5 items in general health perceptions, 4 items in physical role functioning, 3 items in emotional role functioning, 2 items in social role functioning, and 5 items in mental health. The score for each domain will be transformed to a scale from 0 to 100, on which zero corresponds to "worst health status" and 100 to "best health status".
Efficacy-Whole-Organ Magnetic Resonance Imaging Score (WORMS) | Week 24、Week 52、Week 104
  Changes from baseline in Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the target knee.
  MRI performed on the target knee will be used to evaluate the Whole-Organ-MRI Scores (WORMS). The WORMS, diffusion mapping (apparent diffusion coefficient [ADC] and fractional anisotropy [FA]), and T2 map values (it is a value from the worst region for screening visit), will be recorded in the CRF to evaluate the effect on knee cartilage response.
  WORMS are used to evaluate the articular cartilage lesions at three joints, including 14 anatomic compartments as follows (Peterfy et al., 2004)
Efficacy-knee joint space width (JSW) | Week 24、Week 52
  Change from baseline in knee joint space width (JSW) of the target knee. Knee X-ray for knee joint space width (JSW) assessment will be performed on anterior-posterior (AP) view, Rosenberg's view, and axial view of patella 45° (lateral part and medial part). X-ray will be performed for both knees at Screening Visit, while only for the target knee at the other scheduled visits.
Efficacy-synovial fluid | Week 52
  Change from baseline in the synovial fluid analysis of the target knee at Week 52, if the subject's knee is suitable for arthrocentesis per investigator's judgment.
  The volume of synovial fluid aspiration will be determined by the investigator and will be recorded in the CRF. The appearance, white blood cell count (WBC), red blood cell count (RBC), lymphocytes, monocytes, and neutrophils will be examined.
Efficacy-rescue medication | Week 4 to Week 52 、Week 24 to Week 104
  Percentage of subjects using the rescue medication(s) during Visit 3 to Visit 7 and Visit 3 to Visit 8.
  Subjects are allowed to take acetaminophen and/or designated NSAID as rescue medicine to reduce the pain when needed. The acceptable NSAIDs are Etoricoxib and Celebrex. The maximum oral doses for acetaminophen, Etoricoxib, and Celebrex are ≤ 2000 mg/day, ≤ 120 mg/day, and 200 mg/day, respectively, while the topical use of these three rescue medications is allowed at any dose levels.
Safety-AE/SAE based on NCI-CTCAE v5.0 | Week 4、Week 12、Week 24、Week 36、Week 52、Week 104
  The incidence of adverse event (AE)/serious adverse event (SAE). All AEs will be assessed for severity by the investigator based on NCI-CTCAE v5.0. Further, the investigator will judge if the AE is IP-related. Refer to Section 8.4 for details of AE definition and reporting.
Safety-vital signs | Week 4、Week 12、Week 24、Week 36、Week 52、Week 104
  Changes from baseline at each post-treatment visit in vital signs. Vital signs measurement will consist of systolic/diastolic blood pressure, respiratory rate, pulse rate, and body temperature. Respiratory rate, pulse rate, and blood pressure (systolic/diastolic) will be obtained after the subject has been at rest for at least 5 minutes in a sitting position. Vital signs will be performed before and one hour after the Chondrochymal® or HA administration.
Safety-laboratory examination | Week 4、Week 12、Week 24、Week 36、Week 52、Week 104
  Changes from baseline at each post-treatment visit in laboratory examination.
  Laboratory tests to be measured in this study will consist of the following:
  * Hematology: WBC, RBC, hemoglobin, hematocrit, platelet, neutrophils, lymphocytes, monocytes, eosinophils, basophils, prothrombin time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR, Screening only).
  * Biochemistry: blood urea nitrogen (BUN), creatinine, albumin, total protein, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, C-reactive protein (CRP), and estimated glomerular filtration rate (eGFR) calculated by the Modification of Diet in Renal Disease (MDRD) equation (screening only).
Safety-physical examination | Week 4、Week 12、Week 24、Week 36、Week 52、Week 104
  Abnormal findings in physical examination. Physical examination conducted in this study will include the following items: general appearance, skin, eyes, ears, nose, throat, head and neck, heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological system, and other body systems if applicable for describing the status of the subject's health.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - Taipei Municipal Wangfang Hospital (Managed by Taipei Medical University), Taipei, Wenshan District

IPD SHARING:
Plan to Share IPD: No